CLINICAL TRIAL: NCT02992314
Title: Determination of the Safety and Effectiveness of an Oral Rinse in the Reduction of Medication Associated Metallic Taste
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: You First Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MQ-101-16
Record Dates: First submitted 2016-11-30; First posted 2016-12-14 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Medication Associated Metallic Taste , Dysgeusia
MeSH Terms: conditions — Dysgeusia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Metaqil™ Oral Rinse (Experimental): In this arm the test article, Metaqil ™ oral rinse, a proprietary formulation of agents including Monk fruit extract, which can minimize the metallic taste in the mouth caused by the patient's medications.
  Subjects rinse twice a day with 10 mL of the oral rinse for 30 seconds for 30 days.
  They will note, in the daily oral hygiene diary, the date and time of brushing and rinsing.
  Interventions: Device: Metaqil™ Oral Rinse
- Placebo Oral Rinse (Placebo Comparator): This arm will use a placebo with out the active ingredients same way the experimental arm do.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Metaqil™ Oral Rinse — Metaqil™ is a proprietary formulation of GRAS ingradients
  Arms: Metaqil™ Oral Rinse
Device: Placebo — Placebo formulation with out the active ingredients
  Arms: Placebo Oral Rinse

SUMMARY:
Patients taking chemotherapeutic agents often do not comply well with their dosing regiment since many of these medications cause a metallic taste in the mouth. The primary intent is to determine the effectiveness of the oral rinse in reducing the metallic taste in the mouth associated with various chemotherapeutic agents. This clinical study a randomized, double-blind, single-treatment, parallel design with a placebo as the control. The duration of the trial will be 1 month.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has read, signed and received a copy of the Informed Consent and HIPAA authorization prior to study initiation.
2. Subject is able to follow verbal and/or written instructions, perform oral hygiene procedures and return to the test facility for specified study examinations.
3. Subject is between the ages of 18 and 75 years inclusive.
4. Subject will not have professional cleaning during the 3-month trial.
5. Subject has no history of allergy to personal care consumer products, or their ingredients, relevant to any ingredient in the test drug, as determined by the Principal Investigator.
6. Subject has a minimum of 16 natural teeth and a complaint of moderate to severe medication associated metallic taste.
7. Subject agrees to refrain from the use of any oral rinse, toothpaste or dentifrice other than the Colgate® Cavity Protection Fluoride toothpaste and study rinse provided on Visit 1 for the duration of the study.
8. Subject agrees to refrain from the use of other oral care products not supplied by the study center
9. Subject agrees to be compliant with study procedures.
10. Females of childbearing potential agree to use an adequate method of birth control and agree to pregnancy testing at the first and second visit.

Exclusion Criteria:

1. Subject has a condition that requires prophylactic antibiotics for dental examinations and treatments (e.g., has a history of valvular heart disease or a recently placed prosthetic joint).
2. Subject has disqualifying acute or chronic medical illness as judged by the Principal Investigator.
3. Subject is currently taking phenytoin, cyclosporin, nifedipine or any other drug that has been shown to cause gingival enlargement or affect the gingivae.
4. Subject has taken antibiotics, steroids, or non-steroidal anti-inflammatory drugs (e.g., aspirin, ibuprofen) within one week prior to baseline examination. Subjects taking long-term aspirin (81 mg/day) may be included in the trial, but subjects taking a larger dose will be excluded. Subjects taking blood thinners such as Coumadin (warfarin), Lovenox, or Plavix will be excluded.
5. Subject is pregnant (based on pregnancy result) or lactating.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Relief of medication associated metallic taste | 4 weeks
  Have patient complete a VAS ( visual analogue scale) scoring of the degree of metallic taste in the mouth as well as a VAS scoring of the amount of relief of the metallic taste..

SECONDARY OUTCOMES:
Safety evaluation of the test Oral Rinse | 4 Weeks
  Evaluate extra- and intra- oral areas for any mucosal irritation or pathology.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontics and Endodontics,School of Dental Medicine, University at Buffalo, SUNY, Buffalo, New York, United States